CLINICAL TRIAL: NCT01882829
Title: Targeting the NMDA Glutamate Receptor as Novel Antidepressant Strategy: A Pilot Clinical Trial of Nuedexta in Treatment-Resistant Major Depression
Brief Title: Nuedexta in Treatment-Resistant Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James Murrough (Other)
Responsible Party: Sponsor-Investigator, James Murrough, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-0389; IF1463152
Record Dates: First submitted 2013-06-14; First posted 2013-06-20 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Major Depressive Disorder; Treatment Resistant
Keywords: depression; major depressive disorder; treatment resistant; Nuedexta; dextromethorphan; antidepressant; glutamate; NMDA receptor
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nuedexta (dextromethorphan/quinidine) (Experimental): 45/10 mg every 12 hours x 8 weeks
  Interventions: Drug: dextromethorphan/quinidine

INTERVENTIONS:
Drug: dextromethorphan/quinidine — up to 45/10 mg every 12 hours in patients with TRD with a short 7 day tapering period in which subjects are tapered off 45/10 mg dose from twice a day to once daily for an additional 7 days at post 8-week treatment period to minimize the potential for discontinuation effects
  Other Names: Nuedexta

SUMMARY:
There is an urgent need, therefore, to identify well-tolerated, orally available compounds that target the NMDA receptor as a novel treatment approach for TRD. The current project aims to test the safety, tolerability and efficacy of Nuedexta - containing the NMDA antagonist dextromethorphan.

DETAILED DESCRIPTION:
Approximately one-third of patients with major depressive disorder do not achieve adequate symptom control despite a series of multiple treatment trials with currently available antidepressant medication (for example a serotonin-selective reuptake inhibitor). This group of patients - representing treatment-resistant depression (TRD) - accounts for an alarmingly high public health burden and signifies a critical area of need in pharmaceutical treatment development. While current treatments are slow to act and only partially effective, new basic and clinical research focusing on the glutamate system is yielding promising new avenues for novel drug discovery. Ketamine - a glutamate N-methyl-d-aspartate (NMDA) receptor antagonist - has now been demonstrated in several studies to bring about a rapid and robust antidepressant effect, even in patients suffering from TRD. Ketamine is limited as a treatment for TRD by the need for intravenous administration and the potential for untoward medical or psychiatric adverse effects. There is an urgent need, therefore, to identify well-tolerated, orally available compounds that target the NMDA receptor as a novel treatment approach for TRD. The current project aims to test the safety, tolerability and efficacy of Nuedexta - containing the NMDA antagonist dextromethorphan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, 18-65 years of age;
* Current primary Axis I diagnosis of major depressive disorder according to DSM-IV-TR criteria as determined by a psychiatrist and confirmed with the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID);
* Current treatment-resistant depression defined by a history of inadequate response to a minimum of 2 adequate antidepressant treatment trials determined by patient history and chart review and confirmed with the Antidepressant Treatment History Form (ATHF);
* Participants must be willing to discontinue treatment with concomitant medications that are disallowed by the study protocol;
* Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process.

Exclusion Criteria:

* Lifetime diagnosis of schizophrenia or any psychotic disorder, bipolar disorder, pervasive developmental disorders or mental retardation
* Diagnosis of a substance use disorder within the past 1 year ;
* Female participants who are pregnant, nursing, for may become pregnant;
* Any unstable medical illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease); endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease;
* Participants with clinically significant abnormalities of laboratories, physical examination, or ECG;
* Prolonged QT interval, congenital long QT syndrome, history suggestive of torsades de pointes, or heart failure;
* Complete atrioventricular (AV) block without implanted pacemaker, or patients at high risk of complete AV block
* Participants with a history of quinidine, quinine or mefloquine-induced thrombocytopenia, hepatitis, or other hypersensitivity reactions;
* Participants judged to be at serious suicidal risk by the PI;
* Concomitant use with quinidine, quinine, or mefloquine;
* Participants with known hypersensitivity to dextromethorphan;
* Use with an MAOI or within 14 days of stopping an MAOI;
* Concomitant use with drugs that prolong QT interval and are metabolized by CYP2D6

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Murrough JW, Wade E, Sayed S, Ahle G, Kiraly DD, Welch A, Collins KA, Soleimani L, Iosifescu DV, Charney DS. Dextromethorphan/quinidine pharmacotherapy in patients with treatment resistant depression: A proof of concept clinical trial. J Affect Disord. 2017 Aug 15;218:277-283. doi: 10.1016/j.jad.2017.04.072. Epub 2017 Apr 29. PMID 28478356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from October 2013 to December 2015
Period: Overall Study
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Started | 20
Completed | 14
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Nuedexta (Dextromethorphan/Quinidine): up to 45/10 mg every 12 hours x 8 weeks then once a day for 1 week
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Montgomery-Asberg Depression Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The MADRS-S has 10-items which are based on mood symptoms over the past 7 days. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
  units on a scale | 32.5 (3.9)
Clinical Global Impression - Severity (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  units on a scale | 4.5 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: The Montgomery-Asberg Depression Rating Scale is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Each of the 10 items is s scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression). Primary outcome is change in MADRS at Visit 6 (Week 10). Higher values represent a worse outcome.
Time Frame: At baseline and visit 6 (week 10)
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 20
change in units on a scale | -13.0 (11.5)

2. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire Short Form
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire Short Form is a reliable and valid self-report measure designed to obtain sensitive measures of the degree of enjoyment and satisfaction experienced by individuals. The raw total score ranges from 14 to 70. Higher scores reflect better oucomes.
Time Frame: At baseline and Visit 6 (week 10)
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 20
change in units on a scale | 0.1 (0.2)

3. Secondary Outcome: Range of Impaired Functioning Tool
Description: The Range of Impaired Functioning Tool a brief scale for assessing functional impairment related to medical or psychiatric illness and has been demonstrated to possess good psychometric properties. The LIFE-RIFT has a total score and individual domain scores for the following areas of functioning: household duties, work, recreation, relationships with family, relationships with friends, schoolwork, and global life satisfaction (the satisfaction item is patient rated).
  Higher scores indicate poorer functioning; scores ≥2 reflect impaired functioning in that domain. Results are reported for the total sum with full range from 3 (no impairment) to 60 (severe impairment), which is based on all individual domain scores.
Time Frame: At baseline and Visit 6 (week 10)
Population: missing data on 2 participants
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 18
change in units on a scale | -3.7 (4.1)

4. Secondary Outcome: Sheehan Disability Scale
Description: The Sheehan Disability Scale (SDS) is a self-rated scale which assesses illness-related disability in three areas of functioning: work, social and family. The SDS assess disability or functional impairment across three domains: work/school, social life/leisure activities and family life/home responsibilities. Each domain is scored from 0 (not at all) to 10 (very severely). The three domains can be summarized to evaluate global functional impairment by adding the scores of each of the three domains, resulting in global SDS score ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: At baseline and Visit 6 (week 10)
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 20
change in units on a scale | -4.3 (7.4)

5. Secondary Outcome: Patient Rated Inventory of Side Effects (PRISE)
Description: Frequency of observed adverse events over the study treatment period as captured by the PRISE. The Patient Rated Inventory of Side Effects (PRISE) assesses the presence of treatment side effects in nine organ/function systems (gastrointestinal, nervous system, heart, eyes/ears, skin, genital/urinary, sleep, sexual functioning, and other).
Time Frame: up to 12 weeks
Measure: Number; unit: events
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 20
events | 25

6. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a comprehensive, semi-structured interview measure that uniquely measures the full spectrum of suicidality including passive and active suicidal ideation, suicidal intent as well as suicidal behaviors. Full range from 0 (low intensity suicidal ideation to 9 (high intensity suicidal ideation).
Time Frame: up to 12 weeks
Population: missing data on one participant
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 19
change in units on a scale | 0.1 (0.5)

7. Secondary Outcome: Quick Inventory of Depressive Symptomatology, Self Report (QIDS-SR)
Description: The Quick Inventory of Depressive Symptomatology, Self Report (QIDS-SR) is a 16-item self rated instrument designed to assess the severity of depressive symptoms (30). The 16 items cover the nine symptom domains of major depression, and are rated on a scale of 0-3. Total score ranges from 0 to 27, with ranges of 0-5 (normal), 6-10 (mild), 11-15 (moderate), 16-20 (moderate to severe), and 21+ (severe).
Time Frame: up to 12 weeks
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 20
change in units on a scale | -5.9 (6.6)

8. Secondary Outcome: Clinical Global Impression (CGI) Scale
Description: The Clinical Global Impression (CGI) scale assesses overall treatment response in psychiatric patients and has good reliability and validity metrics. The administration time is 2 minutes. This scale consists of three items: Severity of Illness (item 1); Global Improvement (item 2); and Efficacy Index (item 3). Item 1 is rated on a seven-point scale (1 = normal, 7 = among the most extremely ill patients) as is item 2 (1 = very much improved, 7 = very much worse). Full scale is 1 to 14.
Time Frame: up to 12 weeks
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 20
change in units on a scale | -1.5 (1.3)

9. Secondary Outcome: Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ)
Description: The Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) is a brief scale to measure cognitive and executive dysfunction in mood and anxiety disorders, and possesses good reliability and validity. The Massachusetts General Hospital CPFQ was developed to assess each of the 7 most common complaints of depressed patients reporting fatigue or cognitive/executive problems. The CPFQ consists of 7 questions, each rated on a scale from 1 to 6, with 1 indicating greater than normal functioning, 2 indicating normal functioning and with higher numbers indicating poorer functioning. Total score range from 7 (greater than normal function) to 42 (poor function).
Time Frame: At baseline and Visit 6 (week 10)
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 20
change in units on a scale | -4.1 (6.5)

10. Secondary Outcome: HAM-A
Description: Change in Hamilton Anxiety Rating Scale (HAM-A) score from baseline to Week 10. It consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and >25-30 moderate to severe.
Time Frame: Baseline and Week 10
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 20
change in units on a scale | -5.7 (5.9)

11. Secondary Outcome: Beck Scale for Suicidal Ideation (BSI)
Description: Mean change in Brief Inventory Symptom from baseline to week 10. The BSS is a self-report 19-item scale preceded by five screening items. The BSS and its screening items are intended to assess a patient's thoughts, plans and intent to commit suicide. All 24 items are rated on a three-point scale (0 to 2). In this study, scores from the five screening items were included in the overall score. Therefore, total scores could range from 0 to 48, with higher scores reflecting more severe symptoms.
Time Frame: Baseline and Week 10
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
Number analyzed (Participants) | 20
change in units on a scale | -2.5 (5.1)

ADVERSE EVENTS:
Arm/Group | Nuedexta (Dextromethorphan/Quinidine)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nuedexta (Dextromethorphan/Quinidine) (N=20)
Insomnia (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nuedexta (Dextromethorphan/Quinidine) (N=20)
Palpitations (Cardiac disorders) | 1
Vision blurred (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Decreased appetitie (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Sedation (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Mental Status Changes (Psychiatric disorders) | 1
Restlesness (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes